CLINICAL TRIAL: NCT05612022
Title: Acoustic Analysis of Blood Flow-emitted Sounds to Detect Vascular Complications in Arteriovenous Fistulae and Grafts for Hemodialysis
Brief Title: Acoustic Analysis of VA Sounds
Acronym: VAsound
Status: Recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: VAsound
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: End Stage Renal Disease; Hemodialysis Access Failure
Keywords: AVF; AVG; VA sounds; acoustic analysis; VA remodelling; Doppler Ultrasound
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1. Patients with AVF as first line HD access option.: 24 consecutive patients in need of AVF enrolled at the Nephrology and Dialysis unit of the ASST-Papa Giovanni XXIII of Bergamo.
  Interventions: Procedure: AVF creation
- Group 2. Patients with AVG as first line HD access option.: 20 consecutive patients in need of AVG enrolled at the Nephrology and Dialysis unit of the ASST-Papa Giovanni XXIII of Bergamo.
  Interventions: Procedure: AVG creation

INTERVENTIONS:
Procedure: AVF creation — AVF is surgically created in the forearm by an anastomosis between a vein and an artery
  Groups: Group 1. Patients with AVF as first line HD access option.
Procedure: AVG creation — Surgery is done using an artificial plastic tube that connects an artery to a vein
  Groups: Group 2. Patients with AVG as first line HD access option.

SUMMARY:
End-stage renal disease (ESRD) is a growing global health problem, strictly connected with progressive ageing population and longer survival of patients living on renal replacement therapy. The majority of ESRD patients is on hemodialysis (HD) treatment. A successful HD procedure requires a functioning vascular access (VA) to provide safe and long-lasting way to connect patient circulation to the artificial kidney. The current recommendation for VA is the native arteriovenous fistula (AVF), surgically created in the forearm by an anastomosis between a vein and an artery. The AVF, despite being the first-choice treatment, is still affected by high non-maturation and early failure rates, requiring in most of the cases, the creation of a new VA. An arteriovenous graft (AVG) is the second choice for a VA. Surgery is done using an artificial plastic tube that connects an artery to a vein. The AVG matures earlier than AVF (2/3 vs 6 weeks), but it is more prone to infections and has lower survival.

It would be important to identify patients at risk of VA failure, but there is currently a lack of adequate strategies for surveillance. A continuous monitoring of the VA function would help in identification of reduced blood flow and VA stenosis, that could be treated by interventional radiologists before AVF or AVG complete closure. Over the years, nurses and nephrologists got used to touch the VA and qualitatively evaluate its vibration, named "thrill", and the sounds emitted by the same using their stethoscope.

The purpose of this study is to assess the feasibility of VA sound recording and analysis and provide preliminary evidence of VA sound clinical validity and utility to assess, monitor and predict vascular remodelling occurring in AVFs and AVGs.

This is a single center prospective observational study involving the acquisition of VA sounds and Doppler US examinations in consenting patients with ESRD.

To reach this goal, two groups of ESRD patients in need of VA surgery to perform HD treatment will be involved:

Group 1. Patients with AVF as first line HD access option.

Group 2. Patients with AVG as first line HD access option.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Patients in HD treatment that need a new VA or patients that entered the pre-dialysis program because of ESRD. In all these cases the treatment of first choice should be the creation of a distal autogenous AVF, the creation of an AVG or the proximalization of an occluded VA.

Exclusion Criteria:

1. Contraindications for the creation of an autogenous AVF, for the AVG creation or the proximalization of a failed VA.
2. Patients who use catheter to perform HD.
3. Patients undergoing peritoneal dialysis.
4. Patients with life expectancy less than 2 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in patients with ESRD enrolled at the Nephrology and Dialysis Department of the ASST Papa Giovanni XXIII (Bergamo, Italy). VA sounds and Doppler US data will be collected.
  The patients of both groups (AVF and AVG) will undergo visit V1 (screening and enrolment). On day 0 they will have the surgery for VA creation (V2). Then the study follow-up visits will be performed:
  * At 7, 14, 28, 42 and 60 days after VA surgery (V3, V4, V5, V6, V7)
  * Once every 3 months from the third month to two years after VA surgery (V8, …, ENDV).
  Patients will be asked to provide consent for the use of their clinical and laboratory data collected during routine clinical practice over 10 years following the end of this study. Refusal to this consent will not prevent from participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Low-high peak ratio (LHPR) | From v3 (day 7) to end visit (month 24): change from previous visit
  Ratio between the amplitude of maximum peak in the range of lowfrequency (100-250 Hz) and the amplitude of the maximum peak at high frequency (500-750 Hz).

SECONDARY OUTCOMES:
Correlation coefficient between LHPR and Blood Flow Volume (BFV) during VA maturation. | From v3 (day 7) to VA maturation (v6, day 42): change from previous visit
  BFV is measured with Doppler ultrasonography (US).
Correlation coefficient between LHPR and Blood Flow Volume (BFV) after VA maturation. | From v7 (day 60) to end visit (month 24): change from previous visit
  BFV is measured with Doppler ultrasonography (US).

CONTACTS AND LOCATIONS:
Locations (1):
- ASST HPG23 Unità di Nefrologia e Dialisi, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: Undecided